CLINICAL TRIAL: NCT04146714
Title: Screening for Excessive Substance Use in the Waiting Room to Encourage Behavior Change Among Young People (YP-HEALTH): a Multi-center Randomized Controlled Trial in Primary Care
Brief Title: Substance Use Screening to Encourage Behavior Change Among Young People in Primary Care
Acronym: YP-HEALTH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dagmar M. Haller (Other)
Responsible Party: Sponsor-Investigator, Prof. Dagmar M. Haller, Professor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YP-HEALTH
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Substance Use; Binge Drinking; Cannabis Use; Adolescent Behavior
MeSH Terms: conditions — Substance-Related Disorders; Binge Drinking; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants: Although they cannot be masked to the content of the intervention (questionnaire), they are only informed that the study is about health behaviours in general and not specifically about substance use. Thus, they are masked as to whether they are in the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substance use screening (Experimental): Participants complete a substance use questionnaire (=intervention).
  Interventions: Other: Substance use questionnaire
- Physical activity screening (Active Comparator): Participants complete a physical activity questionnaire (=control).
  Interventions: Other: Physical activity questionnaire

INTERVENTIONS:
Other: Substance use questionnaire — Screening questionnaire about substance use based on the Detection of Alcohol and Drug Problems in Adolescents (DEP-ADO) survey.
  Arms: Substance use screening
Other: Physical activity questionnaire — Screening questionnaire about physical activity, based on the short version of the International Physical Activity Questionnaire (IPAQ).
  Arms: Physical activity screening

SUMMARY:
This study evaluates whether completing a short screening questionnaire about health behaviours in the waiting room before a primary care consultation decreases excessive substance use in young people aged 14 to 24 years. Young people consulting a primary care physician will randomly receive either a questionnaire about substance use or a questionnaire about physical activity. They will be contacted again 3, 6 and 12 months later and asked to complete a questionnaire about substance use. The proportion of young people with excessive substance use in each group will be compared. The researchers hypothesise that at three months this proportion will be lower in the group of young people having completed the initial questionnaire about substance use when compared to the group having completed the questionnaire about physical activity.

DETAILED DESCRIPTION:
Background: Excessive alcohol and other substance use often begin in adolescence and contribute extensively to the development of non-communicable diseases and lifelong morbidity/mortality. In Switzerland, the prevalence of binge drinking (the most common mode of alcohol excess in adolescence) and other excessive substance use in young people is high, both in the general and in the primary care population. Since most young people visit a primary care physician at least once in any year, primary care offers an ideal context to individualize the preventive messages delivered in the community to favor behavior change.

Primary care physicians are encouraged to screen and provide brief interventions addressing excessive alcohol and other substance use in young people, but a range of barriers such as time constraints and insufficient training limit the implementation of these recommendations. Finding new ways of building on the potential of primary care whilst addressing these barriers is essential.

Several recent trials of brief primary care interventions showed substantial reductions (20% to 30%) in the proportion of participants who were excessive substance users at follow-up but no statistically significant differences between the intervention and control groups. Key authors have hypothesized that this could be due to assessment reactivity, i.e. when pre-intervention assessment itself encourages behavior change and thus serves as an intervention. Indeed, screening in the clinical context could act as an intervention and be as effective as a brief intervention within the consultation. To date this hypothesis has not been explored for young people attending primary care.

Methods: One of our previous trials (PRISM-Ado), and a pilot trial published in 2019, inform the methods of this parallel-group randomized controlled trial in primary care. Advisory panels of primary care physicians and young people contributed to the development of this protocol. Recruitment will take place in primary care practices in the French-speaking part of Switzerland. Young people between the ages of 14 and 24 years consulting for any health problem will be eligible. Up to 840 young people (approx 20 per practice) will be included and randomized to complete two different types of confidential pre-consultation screening surveys: one focusing on the assessment of binge drinking and other substance use (intervention group) and the other on physical activity (control group). Both surveys will include identical additional socio-demographic and health-related questions. The primary care physicians will not automatically have access to the answers provided in the surveys and participants will be free to decide if they wish to disclose them to their physician during the consultation. Follow-up phone interviews will take place at 3, 6 and 12 months. They will be identical for all participants and include all questions from the intervention and control questionnaires. The main outcome at 3 months follow-up will be the proportion of patients reporting binge drinking (≥1 episode) in the past 30 days. Secondary outcomes will include the proportion of young people reporting smoking (≥ 1 cigarette a day), electronic cigarette use (≥ once a day) and/or excessive cannabis use (≥1 joint/week) in the past 30 days. Analysis will be by intention to treat and will take into account clustering of participants within practices.

Expected value of the proposed trial: If our intervention proves effective, it will offer a simple, widely expandable method to encourage behavior change in young people consulting in primary care, thus contributing to a much-needed reduction in the burden of non-communicable diseases in the future. In addition, by providing a quantification of the effect of assessment reactivity per se, our study will provide key information for the design of future trials of interventions addressing substance use in young people attending primary care.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 14 to 24 years consulting at the participating primary care practice for any motive.

Exclusion Criteria:

* Acute illness requiring immediate attention of the physician
* Severe mental health conditions requiring treatment in a specialized setting
* Young person not consulting as a patient at the practice (e.g. accompanying friend or partner)
* Inability to read the trial information in French or to provide independent consent.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reporting one or more episodes of binge drinking in the past 30 days. | 3 months
  Patient self-report on follow-up telephone questionnaire. Binge drinking is defined as the consumption of five or more standard drinks in one occasion.

SECONDARY OUTCOMES:
Proportion of patients reporting smoking one or more cannabis joints per week in the last 30 days. | 3 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting smoking one or more cannabis joints per week in the last 30 days. | 6 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting smoking one or more cannabis joints per week in the last 30 days. | 12 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting smoking at least one cigarette per day in the last 30 days. | 3 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting smoking at least one cigarette per day in the last 30 days. | 6 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting smoking at least one cigarette per day in the last 30 days. | 12 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting electronic cigarette use at least once per day in the last 30 days. | 3 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting electronic cigarette use at least once per day in the last 30 days. | 6 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting electronic cigarette use at least once per day in the last 30 days. | 12 months
  Patient self-report on follow-up telephone questionnaire.
Proportion of patients reporting one or more episodes of binge drinking in the past 30 days. | 6 months
  Patient self-report on follow-up telephone questionnaire. Binge drinking is defined as the consumption of five or more standard drinks in one occasion.
Proportion of patients reporting one or more episodes of binge drinking in the past 30 days. | 12 months
  Patient self-report on follow-up telephone questionnaire. Binge drinking is defined as the consumption of five or more standard drinks in one occasion.

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar M Haller, MD,PhD, Principal Investigator — Faculty of Medicine, University of Geneva
Locations (1):
- University Institute for Primary Care, Faculty of Medicine, University of Geneva, Geneva, Switzerland